CLINICAL TRIAL: NCT02136433
Title: Using Tablets for Upper Extremity Rehabilitation Post Acquired Brain Injury
Acronym: TBL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-13-0125-RK-CTIL
Record Dates: First submitted 2013-09-02; First posted 2014-05-13 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Brain Injury; Stroke
Keywords: Hand; Rehabilitation; Stroke; Brain-injury; Tablet
MeSH Terms: conditions — Brain Injuries; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet - self exercise (Experimental): Existing tablet Apps that encourage finger movement in a fun manner while playing a game will be used. The apps will be taught to the participants and then they will be requested to exercise alone (or with family) everyday for one hour in addition to their regular rehabilitation sessions (Occupational, Physical Therapy, speech).
  The intervention will include 15-20 sessions of 60 minutes of self-training using a tablet.
  Interventions: Device: Tablet - self exercise
- GRASP self exercise (Active Comparator): GRASP (Graded Repetitive Arm Supplementary Program)(Harris et al., 2009)is an arm and hand exercise program developed for individuals with stroke with upper extremity impairments GRASP provides a method for patients to undertake a self-directed arm and hand exercise program.
  The exercises will be taught to the participants and then they will be requested to exercise alone (or with family) everyday for one hour in addition to their regular rehabilitation sessions (Occupational, Physical Therapy, speech).
  The intervention will include 15-20 sessions of 60 minutes of self-training
  Interventions: Other: GRASP self exercise

INTERVENTIONS:
Device: Tablet - self exercise
  Arms: Tablet - self exercise
Other: GRASP self exercise
  Arms: GRASP self exercise

SUMMARY:
The purpose of the study is to test the effectiveness of training using novel tablet applications for hand function, compared to traditional hand exercises. In addition, we aim to examine brain plasticity following treatment with the new tablet applications. We hypothesize that training with a tablet would prove to be more effective than traditional exercises. We expect to observe neuroplastic changes in the brain in patients who practiced finger movements using the tablet.

ELIGIBILITY:
Inclusion Criteria:

* At least one week post Brain injury or stroke
* Partial ability to open and close their hand (fingers)
* Full function of the hands prior to the injury or event
* Intact or Corrected vision
* Cognitively intact or mild impairment

Exclusion Criteria:

* Other neurological conditions besides the brain injury or stroke
* Orthopedic conditions of the upper extremity

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in score of the Nine Hole Peg Test | An average of one week before intervention and one week after intervention
  To assess dexterity of the affected hand. This test is a assesses dexterity and the time to remove and return nine pegs is measured. The Nine Hole Peg Test is a reliable, valid and responsive measure in clients with stroke

SECONDARY OUTCOMES:
The Fugl-Meyer Motor Assessment | An average of one week before intervention and one week after intervention
  To quantify the level of the motor impairment. The participants are required to perform different movements. Each movement is rated 0 (inability to perform) to 2 (full movement). The total score ranges from 0 (no active movements) to 60 points (full movements).
Grip and pinch strength | An average of one week before intervention and one week after intervention
  Assessed by the Jamar dynamometer. This is a valid and reliable way to assess grip and pinch strength of individuals recovering from stroke.
Visual Analogue Scale | An average of one week before intervention and one week after intervention
  Quantifies the perceived level of pain intensity on a scale of 0-10 cm.
The System Usability Scale | An average of one week after intervention
  This questionnaire includes 10 items which provide a global view of subjective assessment of a system's usability.
Change from baseline in score of the Action Research Arm Test | An average of one week before intervention and one week after intervention
  Assesses the functional ability of the upper extremity by grasping and moving objects of different size and weight. It has four subtests; grasp, grip, pinch and gross movement. The total score is out of 57 points.
Self - report compliance | An average of one week after intervention
  Mean self-training time per day.
Satisfaction Questionnaire | An average of one week after intervention
  Developed for the study and will query how much the subjects were satisfied with the self-training intervention they experienced and to what extent they think it can help them to improve their upper extremity function. Responses will be rated on a scale of 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kizony, PhD, Study Chair — Sheba
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Rand D, Zeilig G, Kizony R. Rehab-let: touchscreen tablet for self-training impaired dexterity post stroke: study protocol for a pilot randomized controlled trial. Trials. 2015 Jun 18;16:277. doi: 10.1186/s13063-015-0796-9. PMID 26081864